CLINICAL TRIAL: NCT00896350
Title: Predicting Treatment Response Based on Hypoxia in Head and Neck Cancers Using Non-Invasive Oxygen Sensitive MRI
Brief Title: MRI in Finding Hypoxia in Patients Undergoing Chemo and Radiation for Head and Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCCC-02308; CDR0000637640 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-02811 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BOLD MRI (Experimental): Determine the amount of oxygen supply to tumors.
  Interventions: Drug: Standard Care Chemoradiation

INTERVENTIONS:
Drug: Standard Care Chemoradiation — External beam radiation to the neck and tumor site of head and neck. Concurrent platinum based chemotherapy. External beam "boost" at discretion of treating physician.

SUMMARY:
RATIONALE: Diagnostic procedures, such as functional MRI, may help measure oxygen levels in tumor cells and may help in planning cancer treatment.

PURPOSE: This phase I trial is studying functional MRI to see how well it works in finding hypoxia in patients undergoing chemotherapy and radiation therapy for stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the undertaken oxygen sensitive MRI for the detection of hypoxia in patients with Stage III-IV head and neck cancer.
* Correlate MRI parameters with histology, gene expression, and plasma osteopontin.
* Correlate tumor hypoxia measurements with patient prognosis and treatment response.

OUTLINE:

* Pre-therapy MRI: Patients undergo blood oxygen level dependant (BOLD) contrast MRI on room air breathing over 2 minutes and with oxygen gas over 15 minutes. Patients also undergo MR-spectroscopy over 15 minutes to measure choline and lactate markers, and dynamic contrast MRI with gadolinium contrast over 8 minutes.
* Chemoradiotherapy: Patients receive platinum based chemotherapy every two weeks. Patients also undergo radiation therapy for 6 weeks.
* Post-radiation MRI: Patients undergo MRI as before chemoradiotherapy. Blood and tumor samples are collected at baseline for biomarker analysis associated with tumor progression or response.

After completion of study, patients are followed every 3 months for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck

  * Stage III or IV disease
* Measurable disease
* Scheduled to undergo standard treatment including radiation therapy and chemotherapy
* Participation on study # 092004-010 for tissue procurement

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Serum creatinine ≤ 1.5 OR creatinine clearance ≥ 40
* Body mass index ≤ 34 Kg/m^2
* Not claustrophobic
* No other contraindications to MRI (i.e., implanted pacemaker device)
* Not pregnant or nursing
* Negative pregnancy test
* No allergy to gadolinium

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07-08 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
MRI signal sensitivity to oxygen | 12 weeks
  MRI signal sensitivity to oxygen breathing and delayed contrast-enhancement (DCE)
Tumor shrinkage and blood oxygen association | 12 weeks
  Association between tumor shrinkage and blood oxygen level dependent

SECONDARY OUTCOMES:
Correlate tumor hypoxia with patient prognosis and treatment response | 12 weeks
  Association between tumor hypoxia, patient prognosis, and treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Baran Sumer, MD, Principal Investigator — Simmons Cancer Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States